CLINICAL TRIAL: NCT00938665
Title: Evaluation of a Handheld Event Related Potential (ERP)/Quantitative Electroencephalography (qEEG) System (COGNISION™) as a Useful Cognitive Biomarker for Alzheimer's Disease.
Acronym: COGNISION™
Status: Completed | Type: Observational
Sponsor: Neuronetrix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SRP-1418
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Memory Disorders; Alzheimer Disease; Dementia; Cognitive Impairment; Frontotemporal Dementia
Keywords: Alzheimer; Memory disorder; dementia; cognitive behavioral decline; vascular dementia; front temporal dementia
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease; Dementia; Cognitive Dysfunction; Frontotemporal Dementia; Dementia, Vascular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. These lab tests will be performed from a standard blood draw:
     1. B12
     2. TSH
     3. CRP
     4. ALT
     5. HGB
     6. Hgb1AC
     7. T4
     8. Na
     9. K
     10. Cl
     11. CO2
     12. ApoE
     13. Platelet Count
     14. INR
     15. PT
  2. MRI- INCLUDING VOLUMETRY
  3. CSF 5ML (Optional)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group
  Interventions: Device: COGNISION™ System
- AD Group
  Interventions: Device: COGNISION™ System

INTERVENTIONS:
Device: COGNISION™ System — 30 minute ERP test and 3 minute resting EEG data collected from cognitively healthy and AD to validate ERP and qEEG as useful cognitive biomarkers for AD.

SUMMARY:
The proposed study is designed to evaluate the performance of the COGNISION™ System as a tool to assist physicians in diagnosing Alzheimer's Disease (AD) in real-world clinical settings. The design of this study is guided by two overriding factors: 1) to optimize the performance of the event related potentials (ERP) classifiers, the subjects making up the training sets must be well characterized as to their clinical diagnosis, and 2) all ERP tests must be performed and reproduced in real-world clinical settings.

DETAILED DESCRIPTION:
The study will be :

A. Multi-Center Study:

primary goal of this study will be to evaluate the COGNISION™ Platform across multiple study locations. This will demonstrate an ability to perform tests, collect data, and generate classifications irrespective of variations in testing locations and personnel.

1. 5-8 study sites will be selected with each site being a recognized NIH Center of Excellence for Alzheimer's disease or other nationally recognized Alzheimer's disease research center.
2. Each site will evaluate up to 60 subjects evenly divided between AD patients and age-matched controls (while the prevalence of AD is approximately 2% in the general population, the ratio of AD to normal among those who visit a clinic for memory or cognitive related issues is between 50-60%).
3. Each site will follow the same testing protocols.
4. All test data will be uploaded to the online COGNISION™ database server.

ELIGIBILITY:
Inclusion Criteria:

AD Cohort:

Subjects between 60 and 90 years old meeting NINCDS-ADRDA criteria for probable AD2 and DSM-IV criteria for dementia of the Alzheimer's type3 will be recruited in the AD cohort (MMSE ≥21, ≤26).

Memory complaint by subject and/or study partner SRP-1418 N Page: 8 of 26

Abnormal memory function score on Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised (adjusted for education. Maximum score is 25):

i. < 10 for 16 or more years of education ii. < 6 for 8-15 years of education iii. < 4 for 0-7 years of education Clinical Dementia Rating (CDR) = 0.5, 1.0 or 2.0 Modified Hachinski Ischemic Scale (HIS) ≤ 4 Geriatric Depression Scale (GDS) < 6 For subjects that decide to provide a CSF sample: Platelet count ≥ 100,000/μL, Prothrombin Time (PT) = 11 to 16 seconds, International Normalized Ratio = 0.8 to 1.2 Study partner or caregiver to accompany subject to all scheduled visits Fluent in English Adequate visual acuity to allow neuropsychological testing Adequate auditory acuity to allow neuropsychological and ERP testing Good general health with no additional diseases expected to interfere with the study Willing to undergo neuroimaging and provide blood. The subject may optionally provide a CSF sample by lumbar puncture.

Normal Controls:

Healthy subjects matched for age, gender, and education level will be recruited as normal controls (MMSE ≥ 27).

Normal memory function will be documented by scoring at specific cutoffs on the

Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised:

i. ≥ 10 for 16 or more years of education ii. ≥ 6 for 8-15 years of education iii. ≥ 4 for 0-7 years of education Study partner or caregiver Fluent in English Adequate visual acuity to allow neuropsychological testing Adequate auditory acuity to allow neuropsychological and ERP testing

Exclusion Criteria:

AD Cohort:

Severe or unstable forms of diabetes, heart disease, HIV, drug or alcohol abuse, etc. including severe AD: MMSE ≤20 Platelet count < 100,000/μL, Prothrombin Time (PT) > 16 seconds, International Normalized Ratio > 1.2 (for subjects that choose to provide a CSF sample by lumbar puncture).

Medical or psychiatric disorders that might complicate the assessment of dementia (i.e., mental retardation, alcohol abuse, drug abuse, HIV) A disability that may prevent the subject from completing all study requirements (e.g., blindness, deafness, language difficulty) Recent intake of drugs known to cause major organ system toxicity or CNS alteration (e.g. sedation) Diseases of the dementia type other than AD (i.e., vascular dementia, frontotemporal dementia, Lewy Body Disease, Huntington's disease) Presence of non-MRI compatible implants/devices Prohibited Medications: Warfarin or other anticoagulants (for subjects that choose to provide a CSF sample by lumbar puncture), investigational agents.

Normal Controls:

Severe or unstable forms of diabetes, heart disease, HIV, drug or alcohol abuse, etc.

A disability that may prevent the subject from completing all study requirements (e.g., blindness, deafness, language difficulty) Use of psychoactive drugs (only SSRI's are allowed) Psychiatric disorders (schizophrenia, bipolar, etc.) Depression (GDS > 6) Vascular dementia (HIS > 4) Other dementia (CDR > 0)

Abnormal memory function score on Wechsler Memory Scale -Logical Memory II subscale (delayed Paragraph Recall) from the Wechsler Memory Scale - Revised (the maximum score is 25):

I. < 10 for 16 or more years of education II. < 6 for 8-15 years of education III. < 4 for 0-7 years of education

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects between 60 and 90 years old meeting DSM-IV criteria for dementia of the Alzheimer's type and NINCDS-ADRDA criteria for probable AD will be recruited in the AD cohort. Matched cognitively healthy volunteers will be recruited for the Control group.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Electrophysiological markers of cognitive status | Markers are collected at study visit

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Smith, MD, Principal Investigator — Univeristy of Kentucky; Murali Doraiswamy, MD, Principal Investigator — Duke University; Steven E Arnold, MD, Principal Investigator — University of Pennsylvania; Paul R Solomon, PhD, Principal Investigator — The Memory Clinic, Bennington VT; Bradley S Folley, PhD, Principal Investigator — Norton Healthcare, Louisville KY; Carl Sadowsky, MD, Principal Investigator — Premiere Research Institute, West Palm Beach FL; Andrew E Budson, MD, Principal Investigator — Boston Center for Memory
Locations (7):
- United States (7):
  - Premiere Research Institute, West Palm Beach, Florida
  - University of Kentucky, Lexington, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - Boston Center for Memory, Brookline, Massachusetts
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Memory Clinic, Bennington, Vermont